CLINICAL TRIAL: NCT01626989
Title: Evaluation of the Philips Respironics BiPAP autoSV Devices in Subjects With Sleep Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ST-1007-ASV4-MS
Record Dates: First submitted 2011-05-19; First posted 2012-06-25 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disordered Breathing; Sleep Apnea, Central
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BiPAP auto SV Advanced (Active Comparator): BiPAP auto SV Advanced
  Interventions: Device: BiPAP auto Advanced
- BiPAP auto SV 4 (Experimental): Auto Servo Ventilation Device
  Interventions: Device: BiPAP auto SV4

INTERVENTIONS:
Device: BiPAP auto Advanced — Auto Servo Ventilation Device
  Other Names: BiPAP Auto SV
  Arms: BiPAP auto SV Advanced
Device: BiPAP auto SV4 — Auto Servo Ventilation Device
  Other Names: BiPAP Auto SV
  Arms: BiPAP auto SV 4

SUMMARY:
Comparing two BiPAP autoSV devices in participants with complex sleep apnea and determining if the new device will treat those participants no worse than when compared to its predecessor device.

DETAILED DESCRIPTION:
The use of the BiPAP autoSV4 device in participants with Complex Sleep Apnea Syndrome will treat those participants no worse than when compared to its predecessor device, the BiPAP autoSV Advanced™, with respect to:

• Apnea-Hypopnea Index (AHI)

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80
* Ability to provide consent
* Documentation of medical stability by investigator
* Subjects who currently have been on Positive Airway Pressure (PAP) therapy for ≥ 4 weeks and who previously had a Continuous Positive Airway Pressure (CPAP) titration with CAI ≥ 5.

OR Subjects who currently have been on PAP therapy for ≥ 4 weeks and who had a diagnostic study done, with a CAI ≥ 5, and were prescribed PAP therapy without a CPAP titration.

* Agreement to undergo a full-night, in-lab research CPAP Titration
* Agreement to undergo two full-night, in-lab therapy research Polysomnography (PSG) on BiPAP autoSV devices

Exclusion Criteria:

* Major medical or psychiatric condition that would interfere with the demands of the study, adherence to positive airway pressure, or the ability to complete the study. For example, unstable congestive heart failure, chronic lung disease, neuromuscular disease, daytime hypercapnia, cancer, or renal failure.
* Systolic blood pressure < 80 mm Hg at Baseline Visit.
* Participants in whom PAP therapy is otherwise medically contraindicated.
* Participants who are unwilling to wear CPAP
* Currently prescribed oxygen therapy (as needed, nocturnal, or continuous
* Participants with previously diagnosed respiratory failure or respiratory insufficiency and who are known to have chronically elevated arterial carbon dioxide levels while awake (PaCO2 ≥ 45mmHg).
* Participants who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days.
* Participants with untreated, non-obstructive Sleep Apnea (OSA)/ Complex Sleep Apnea (CSA) sleep disorders, including but not limited to; insomnia, periodic limb movement syndrome, or restless legs syndrome (PLM Arousal Index > 15).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahrokh Javaheri, MD, Principal Investigator — Sleepcare Diagnostics; Paul Wylie, MD, Principal Investigator — Arkansas Center for Sleep Medicine; Mark Goetting, MD, Principal Investigator — Sleep Health
Locations (3):
- United States (3):
  - Arkansas Center for Sleep Medicine, Little Rock, Arkansas
  - Sleep Health, Portage, Michigan
  - Sleepcare Diagnostics, Mason, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Screening Population: All patients that signed consent are considered for the screening population.
- BiPAP Auto SV Advanced First, Then BiPAP Auto SV 4: Participants received the Philips BiPAP Auto SV Advanced for one night, then received the BiPAP Auto SV 4 for one night.
- BiPAP Auto SV 4 First, Then BiPAP Auto SV Advanced: Participants received the Philips BiPAP Auto SV 4 for one night, then received the BiPAP Auto SV Advanced for one night
Period: Screening Period
Arm/Group | Screening Population | BiPAP Auto SV Advanced First, Then BiPAP Auto SV 4 | BiPAP Auto SV 4 First, Then BiPAP Auto SV Advanced
Started | 44 | 0 | 0
Completed | 27 | 0 | 0
Not Completed | 17 | 0 | 0
Not completed — Screen Failure | 15 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: Fist Intervention (Night 1)
Arm/Group | Screening Population | BiPAP Auto SV Advanced First, Then BiPAP Auto SV 4 | BiPAP Auto SV 4 First, Then BiPAP Auto SV Advanced
Started | 0 | 15 | 12
Completed | 0 | 15 | 12
Not Completed | 0 | 0 | 0
Period: Second Intervention (Night 2)
Arm/Group | Screening Population | BiPAP Auto SV Advanced First, Then BiPAP Auto SV 4 | BiPAP Auto SV 4 First, Then BiPAP Auto SV Advanced
Started | 0 | 15 | 12
Completed | 0 | 15 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants that signed consent.
Groups:
- All Study Participants: All study participants that signed consent.
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.71 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 39
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 44
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.3 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index (AHI)
Description: Apnea-Hypopnea Index (AHI) is the number of apneas and hypopneas per hour of sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Continous Positive Airway Pressure Titriation: Baseline Polysomnograph (PSG) to qualify for randomization.
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
events per hour | 38 (31) | 13 (17) | 12 (18)
Statistical Analysis 1: Comparison: BiPAP Auto SV Advanced vs BiPAP Auto SV 4; Test type: Non-Inferiority or Equivalence — Friedman Test comparing all 3 nights; p = .001, nonparametric Wilcoxon Signed Rank test

2. Secondary Outcome: Non Rapid Eye Movement (NREM) and Rapid Eye Movement (REM) Percentage Based on Total Sleep Time (TST) Indices
Description: REM is the period of rapid eye movement sleep, NREM are stages 1, 2, and 3 of sleep, and Total Sleep Time (TST) is the duration of time from "lights out," or bedtime, to the onset of sleep. The amount of actually sleep time in a sleep episode; this time is equal to the total sleep episode less the awake time. TST is the total of all REM and NREM sleep in a sleep episode
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent of TST
Groups:
- Continous Positive Airway Pressure Titriation: Baseline PSG to qualify for randomization.
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
percent of TST
  Stage 1 | 22 (14) | 18 (10) | 17 (10)
  Stage 2 | 61 (14) | 65 (13) | 65 (12)
  Stage 3 | 5 (8) | 4 (6) | 5 (6)
  REM | 11 (9) | 13 (9) | 14 (11)

3. Secondary Outcome: Central Apnea Index(CAI)
Description: Central Apnea Index(CAI) is the number of central apneas divided by the number of hours of sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis. 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
events per hour | 12 (15) | 1 (2) | 1 (3)

4. Secondary Outcome: Obstructive Apnea Index (OAI)
Description: Obstructive Ap8 participants had missing or unscorable data, therefore they are not included in the analysis. nea Index (OAI) is the number of obstructive apneas divided by the number of hours of sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
events per hour | 14 (10) | 1 (2) | 2 (4)

5. Secondary Outcome: Mixed Apnea Index (MAI)
Description: Mixed Apnea Index (MAI) is the number of combination of central and obstructive apneas divided by the number of hours of sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
events per hour | 4 (7) | 0.3 (0.6) | 0.6 (2)

6. Secondary Outcome: Sleep Onset Latency (SOL)
Description: Sleep Onset Latency (SOL) is the amount of time it takes to fall asleep after the lights have been turned off.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
minutes | 16.6 (16.3) | 19.3 (10.1) | 24.3 (20)

7. Secondary Outcome: REM Onset Latency (ROL)
Description: REM Onset Latency (ROL) is defined as the time it takes to get into REM sleep from Sleep Onset.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: REM onset latency is not a standard set of sleep scores analyzed. This is not apart of the analysis, this is in the protocol by error. However the protocol was not amended.
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: Wake After Sleep Onset (WASO) is a statistic used in sleep studies to determine the amount of time a person spends awake, starting from when they first fall asleep to when they become fully awake and do not attempt to go back to sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
minutes | 59.1 (48) | 64.1 (57.6) | 54.2 (29.3)

9. Secondary Outcome: Total Sleep Time (TST)
Description: Total Sleep Time (TST). Total Sleep Time (TST) is the duration of time from "lights out," or bedtime, to waking from sleep. The amount of actually sleep time in a sleep episode; this time is equal to the total sleep episode less the awake time. TST is the total of all REM and NREM sleep in a sleep episode
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
minutes | 354.0 (74.3) | 352.4 (69.2) | 368.1 (64.6)

10. Secondary Outcome: Sleep Efficiency (SE %)
Description: Sleep Efficiency (SE %) is the percentage of time spent asleep while in bed.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent of time asleep
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
percent of time asleep | 82 (13) | 81 (12) | 82 (8)

11. Secondary Outcome: Wake (W), Stages N1,N2,N3 (NREM), and REM (R) Sleep
Description: Wake (W), Stages N1,N2,N3 (NREM), and REM (R) sleep. REM is the period of rapid eye movement sleep, NREM are stages 1, 2, and 3 of sleep, and Wake (W) is the duration of time from "lights out," or bedtime, to the onset of sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: Data was not analyzed as number of minutes, as minutes is not a meaningful measurement. It is best measured respective to % TST in outcome measure 2. This was included in the protocol in error and the protocol was not amended.
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Arousal Index
Description: Arousal Index is the number of arousals and awakenings is registered in the study, and reported as a total number and as a frequency per hour of sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
events per hour | 22 (12) | 16 (7) | 16 (8)

13. Secondary Outcome: Nocturnal Oxygenation
Description: Nocturnal oxygenation measured by continuous pulse oximetry during sleep study.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent oxygen saturation
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
percent oxygen saturation | 82 (7) | 86 (4) | 84 (5)

14. Secondary Outcome: Hypopnea Index (HI)
Description: Hypopnea Index (HI) is the number of hypopneas divided by number of hours of sleep.
Time Frame: Baseline, and 2 nights (1 night for each intervention)
Population: 8 participants had missing or unscorable data, therefore they are not included in the analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Continous Positive Airway Pressure Titriation | BiPAP Auto SV Advanced | BiPAP Auto SV 4
Number analyzed (Participants) | 19 | 19 | 19
events per hour | 9 (9) | 11 (15) | 8 (11)

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- All Participants: All Study participants that were consented to the study.
- BiPAP Auto SV Advanced: All participants that received the Philips BiPAP Auto SV Advanced.
- BiPAP Auto SV 4: All participants that received the Philips BiPAP Auto SV 4.
Arm/Group | All Participants | BiPAP Auto SV Advanced | BiPAP Auto SV 4
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/44 | 0/27 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=44) | BiPAP Auto SV Advanced (N=27) | BiPAP Auto SV 4 (N=27)
Stents (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No